CLINICAL TRIAL: NCT03937739
Title: Nutritional Status and Constipation Scoring for Inguinal Hernia Patients; A Case-Control Study.
Brief Title: Nutrition and Constipation at Inguinal Hernia Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cemile Idiz, Principal Investigator, Istanbul University
Other Study IDs: Hernia nutrition
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Nutrition; Constipation; Inguinal Hernia
Keywords: Nutrition; Constipation; Hernia
MeSH Terms: conditions — Constipation; Hernia, Inguinal; Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Case group,: The patients who admitted to the general surgery for operation with inguinal hernia were the case group of this study.
  Interventions: Other: Nutritional and constipation questionnaire
- Group 2: Control group,: The patients who were admitted to the same hospital with such as eye, ear/nose/throat, dermatologic diseases or elective surgeries and did not have any inguinal hernia complaints, constipation and other chronic disease which could increase the intra abdominal pressure selected as control group.
  Interventions: Other: Nutritional and constipation questionnaire

INTERVENTIONS:
Other: Nutritional and constipation questionnaire — Alcohol and smoking habits, daily activity, frequency of food consumption and the constipation scoring according to Agachan et all. were examined using questionnaire

SUMMARY:
There are lots of inguinal hernia risk factors determined in the literature. But the relationship between nutritional status and inguinal hernia were not examined yet. In this study the investigators evaluated the constipation scale and food consumption of the inguinal hernia patients. This Case-Control study was performed between March 2018- March 2019. The patients who admitted for operation with inguinal hernia were the case group (n:115) and the patients who were admitted to the same hospital without inguinal hernia were control group (n:88). The age, body mass index, alcohol and smoking habits, daily activity, frequency of food consumption and the Wexner constipation scoring were examined using questionnaire were noted.

DETAILED DESCRIPTION:
Inguinal hernia is the most common type of abdominal wall hernias and the prevalence is estimated as 5-10% in United States. Although many risk factors have been defined for inguinal hernia, family history of inguinal hernia has been reported to be one of the most important factors. In addition to this, advanced age, male gender, smoking, chronic cough causing intraabdominal pressure increase, and chronic constipation are the risk factors. The hernias may recur according to the causes they originate from the reasons they originate in the early or late period after treatment.In this study, constipation and nutritional status of inguinal hernia patients were evaluated and it was aimed to examine the relationship between inguinal hernia and nutrition which has not been previously evaluated in the literature.

This Case-Control study was performed between March 2018- March 2019. The patients who admitted to the general surgery for operation with inguinal hernia were the case group of this study (n:115). Also, the patients who were admitted to the same hospital with such as eye, ear/nose/throat, dermatologic diseases or elective surgeries and did not have any inguinal hernia complaints, constipation and other chronic disease which could increase the intra abdominal pressure selected as control group (n:88).

Written informed consent was obtained from each participant. The numbers of cases and controls were matched based gender and age in each group. The age, gender, body mass index, alcohol and smoking habits, daily activity, frequency of food consumption and the constipation scoring according to Wexner constipation scoring were examined using questionnaire. The demographic data, nutritional status and the constipation scores were compared among individuals to identify differences between these two groups.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Inguinal Hernia

Exclusion Criteria:

* Cancer
* Pregnancy
* Chronic liver diseases
* Previous abdominal surgery history
* Femoral hernia
* Bilateral inguinal hernia
* Weight loss above the 20% of the body weight in the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who admitted to the general surgery for operation with inguinal hernia were the case group of this study. Also, the patients who were admitted to the same hospital with such as eye, ear/nose/throat, dermatologic diseases or elective surgeries and did not have any inguinal hernia complaints, constipation and other chronic disease which could increase the intra abdominal pressure selected as control group.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Nutritional frequency | 1 week
  Food consumption questionnaire with;
  Daily cheese consumption (gram) Daily red meat consumption (gram) Daily chicken consumption (gram) Daily fish consumption (gram) Daily salami- sausage consumption (gram) Daily giblets (Liver, kidney etc.) consumption (gram) Daily egg consumption (gram) Daily nuts consumption (gram) Daily legumes consumption (gram) Daily bread consumption (gram) Daily rice-pasta consumption (gram) Daily vegetable consumption (gram) Daily fruit consumption (gram) Daily fastfood consumption (gram)
Physical activity | 1 week
  Regular physical activity (minute/week)
Smoking and alcohol use | 1 week
  Number of daily cigarette usage Glass of daily alcohol use

SECONDARY OUTCOMES:
Constipation scoring | 1 week
  Constipation scoring according to Wexner constipation scale with a 8 question questionnaire.
  First seven questions have 0 to 4 point and the last question has 0 to 2 point in the scoring system. All of these points summed and the minimum and maximum total score is 0 to 30. In this scoring system total score which is above 15 point is significant for constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Idiz, Ph.D, Study Director — Itanbul University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul
  - Istanbul Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
If any researcher want to use our data for metaanalysis we can share.

REFERENCES:
- [Result] Dabbas N, Adams K, Pearson K, Royle G. Frequency of abdominal wall hernias: is classical teaching out of date? JRSM Short Rep. 2011 Jan 19;2(1):5. doi: 10.1258/shorts.2010.010071. PMID 21286228
- [Result] Burcharth J, Pommergaard HC, Rosenberg J. The inheritance of groin hernia: a systematic review. Hernia. 2013 Apr;17(2):183-9. doi: 10.1007/s10029-013-1060-4. Epub 2013 Feb 20. PMID 23423330
- [Result] Kartal A, Yalcin M, Citgez B, Uzunkoy A. The effect of chronic constipation on the development of inguinal herniation. Hernia. 2017 Aug;21(4):531-535. doi: 10.1007/s10029-017-1604-0. Epub 2017 Apr 9. PMID 28393306
- See also: Nutritional suggestions for hernia patients — https://www.niddk.nih.gov/health-information/digestive-diseases/inguinal-hernia.